CLINICAL TRIAL: NCT00205361
Title: Respiratory Tract IgA Levels in Anesthetized Patients Undergoing Elective Surgical Procedures
Brief Title: Airway IgA: Respiratory Tract IgA Levels in Anesthetized Patients Undergoing Elective Surgical Procedures
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-027
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Healthy; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: well-nourished
- 2: malnourished

SUMMARY:
The purpose of the study is to determine the variability of airway IgA levels in anesthetized, well-nourished and malnourished patients undergoing elective general surgical procedures and the effect of gender and race on this baseline variable. The hypothesis is that airway IgA levels are lower in malnourished than in well-nourished patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery via general anesthesia

Exclusion Criteria:

* Patients with a history of asthma or documented airway irritability
* Patients who have undergone previous pulmonary resection
* Patients receiving cardiac medications for arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2002-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kudsk, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States